CLINICAL TRIAL: NCT01190579
Title: Multicenter Evaluation of Coronary Dual Source CT Angiography in Patients With Intermediate Risk of Coronary Artery Stenoses
Brief Title: Dual Source CT Angiography for Detection of Coronary Artery Stenoses
Acronym: MEDIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Siemens Medical Solutions (Industry); Bayer (Industry)
Responsible Party: Stephan Achenbach, University of Erlangen-Nürnberg Medical School
Other Study IDs: MEDIC
Record Dates: First submitted 2010-08-20; First posted 2010-08-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Chest Pain; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The trial will investigate the accuracy of Dual Source CT coronary angiography to detect coronary artery stenoses in patients with chest pain who have, based on clinical criteria, an intermediate likelihood for the presence of coronary artery stenoses. No beta blockers will be used to lower the heart rate for the examination. The hypothesis is that Dual Source CT will allow the detection of vessels with at least one coronary artery stenosis with a sensitivity of more than 90%.

ELIGIBILITY:
Inclusion Criteria:

* suspected coronary artery disease
* chest Pain
* intermediate likelihood of coronary stenoses
* planned invasive coronary angiography
* age 30 to 80 years

Exclusion Criteria:

* non sinus rhythm
* contrast allergy
* renal failure
* unstable clinical condition
* previous coronary revascularization
* calcium score exceeding 800
* inability to perform 10 second breathhold
* possible pregnancy
* metformin medication that cannot be interrupted
* inability to establish antecubital iv access

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chest Pain and an Intermdiate Likelihood for Coronary Artery Stenoses
Sampling Method: Non-Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy for the detection of coronary artery stenoses | 72 hours
  Invasive coronary angiography will be preformed within 72 hours to verify coronary CT angiography results.

SECONDARY OUTCOMES:
Safety of Ultravist 370 and Ultravist 300 for coronary CT angiography | 1 hour
  Patients will be monitored for one hour after injection of Ultravist 370 and Ultravist 300 intravenously to assess safety and detect side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Achenbach, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (8):
- Vejle Medical Center, Vejle, Denmark
- Germany (4):
  - University of Erlangen, Erlangen
  - Roentgenpraxis Hamburg, Hamburg
  - Klinikum Grosshadern, Munich
  - Deutsches Herzzentrum Muenchen, München
- Ravi Bathina, Hyderabad, India
- Cardiovascular Institute, Monterrey, Mexico
- Tan Tok Seng Hospital, Singapore, Singapore